CLINICAL TRIAL: NCT05955118
Title: Hydrus Microstent as a Quality of Life Consideration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: InSight Vision Center Medical Group, Inc (Other)
Responsible Party: Principal Investigator, Eric Poulsen, Ophthalmologist, InSight Vision Center Medical Group, Inc
Other Study IDs: HQoL-23
Record Dates: First submitted 2023-05-25; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Open Angle Glaucoma: Subjects with mild to moderate open angle glaucoma undergoing bilateral combined cataract surgery & Hydrus Microstent implantation.
  Interventions: Device: Hydrus Microstent

INTERVENTIONS:
Device: Hydrus Microstent — Hydrus Microstent placed at the time of cataract surgery

SUMMARY:
The study aims to identify if Hydrus microstent implantation in patients with open angle glaucoma (OAG) at the time of cataract surgery improves quality of life for patients and explore what quality of life factors motivate patients.

DETAILED DESCRIPTION:
Prospective, interventional single arm study of patient-reported outcomes (PRO) via GSS with pre and post ocular surface disease assessment in subjects undergoing bilateral phaco and Hydrus implantation; Study will also explore other QOL factors that may motivate patients to accept Hydrus via Glauc-QOL36 and customized questions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate open angle glaucoma as defined by with visually significant age-related cataract undergoing uncomplicated cataract surgery and Hydrus Microstent
* Current treatment with one or more ocular hypotensive medication
* Corneal thickness between 470 to 610µm
* Potential of good best corrected visual acuity at distance in the investigator's judgement of at least 0.1 LogMAR (20/25) postoperatively

Exclusion Criteria:

* Clinical diagnosis of secondary glaucoma (traumatic, neovascular, mixed-mechanism, uveitic glaucoma)
* corneal opacity or angle abnormalities that make visualizing the angle difficult
* Past ocular surgery
* History of ocular, systemic medications, or systemic diseases/co-morbidities that significantly impact on quality of life or vision (e.g. advanced macular degeneration, autoimmune diseases, mental illness/depression, uncontrolled systemic disease on polypharmacy)
* Severe dry eye requiring secretagogues, serum eyedrops, topical corticosteroids, amniotic membrane grafts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with mild to moderate OAG undergoing bilateral combined cataract surgery & Hydrus Microstent implantation
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Glaucoma Symptom Score (GSS) Score | 3 months
  GSS is a cross-sectional study of symptoms, functional impairment, and vision-targeted health-related quality of life among persons with glaucoma, scored 0-100, with a higher score being more favorable (ie fewer adverse symptoms).

SECONDARY OUTCOMES:
Number of Medication Reduction for Glaucoma | 3 months
  The number of glaucoma medications used before the intervention are compared to the number used after.
Ocular surface disease (OSD) assessment | 3 months
  The Oxford Grading System is used to grade the amount of corneal and conjunctival fluorescein staining, scored 0 (none) to V.

CONTACTS AND LOCATIONS:
Locations (1):
- Terri Smith, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Journal publication. Congress presentation.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT05955118/ICF_000.pdf